CLINICAL TRIAL: NCT06750770
Title: Development and Validation of a Clinical Risk Prediction Model for Early Acute Kidney Injury After Liver Transplantation
Brief Title: Development and Validation of a Clinical Risk Prediction Model for Early Acute Kidney Injury Within 48 Hours After Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 22216-4-01
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Acute Kidney Injury; Liver Transplantation; Model
Keywords: acute kidney injury, liver transplantation, model, validation
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AKI group: Participants who were diagnosed acute kidney injury(AKI)
  Interventions: Diagnostic Test: KDIGO CRITERIA
- Non-AKI group: Participants who were not diagnosed AKI
  Interventions: Diagnostic Test: KDIGO CRITERIA

INTERVENTIONS:
Diagnostic Test: KDIGO CRITERIA — 2012 KDIGO DIAGNOSTIC CRITERIA

SUMMARY:
Acute kidney injury (AKI) is a common complication after liver transplantation, with an incidence of 12.7-95%. The occurrence of acute kidney injury after transplantation is related to the poor prognosis of patients, which significantly increases the length of hospital stay, hospitalization costs and mortality of patients. Early recognition of acute kidney injury after transplantation is of great significance. Therefore, by collecting preoperative and intraoperative variables, this study intends to establish and verify a clinical risk prediction model for early AKI after liver transplantation, in order to provide clinicians with a visual prediction tool to identify patients with high risk of early AKI after liver transplantation immediately after the operation, so as to start clinical intervention as soon as possible and improve the prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent liver transplantation in Beijing Tsinghua Changgung Hospital.

Exclusion Criteria:

* (1) under 18 years of age (2) post-renal transplant (3) liver combined with other organ transplants (4) preoperative requirement for renal replacement therapy (RRT) (5) patients with second or multiple liver transplants (6) preoperative estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m2, and (7) patients with severe illness leading to termination of surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion criteria for our study comprised consecutive patients undergoing liver transplantation at Tsinghua University Beijing Changgung Hospital from January 1, 2018, to October 15, 2022. Exclusion criteria were as follows: (1) under 18 years of age (2) post-renal transplant (3) liver combined with other organ transplants (4) preoperative requirement for renal replacement therapy (RRT) (5) patients with second or multiple liver transplants (6) preoperative estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m2, and (7) patients with severe illness leading to termination of surgery.
Sampling Method: Probability Sample
Enrollment: 453 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
KDIGO criteria (Kidney Disease: Improving Global Outcomes) used to evaluate postoperative AKI in liver transplant patients. | 48 hours post-surgery
  Diagnosed according to 2012 KDIGO criteria: serum creatinine rise ≥50% or ≥26.5 µmol/L within 48 hours post-surgery. Baseline creatinine was the most recent preoperative value, with kidney function assessed by eGFR.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tsinghua Changgung Hospital, Beijing, Province, China

IPD SHARING:
Plan to Share IPD: No